CLINICAL TRIAL: NCT06855537
Title: Randomized Controlled Study on the Effectiveness of Interventional Therapy for Non-Flow-Limiting Vulnerable Plaques
Brief Title: Effectiveness of Interventional Therapy for Non-Flow-Limiting Vulnerable Plaques
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaofan Wu, MD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-04
Record Dates: First submitted 2025-01-13; First posted 2025-03-04 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Coronary Arterial Disease (CAD); Vulnerable Coronary Plaques; Thin-cap fIbroatheroma; Acute Coronary Syndromes (ACS)
Keywords: Optical Coherence Tomography (OCT); Percutaneous Coronary Intervention (PCI); Randomized Controlled Trial (RCT); Optimal Medical Therapy; Drug Eluting Stent (DES); Quantitative Flow Ratio (QFR); Acute Coronary Syndromes (ACS); Vulnerable Coronary Plaques
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PCI+OMT (Experimental): PCI plus guideline-recommended optimal medical therapy (including intensive lipid-lowering therapy [LDL<1.4mmol/l and decreased by 50% compared to the baseline]).
  Interventions: Procedure: PCI strategy; Drug: OMT strategy
- OMT (Active Comparator): Guideline-recommended optimal medical therapy (including intensive lipid-lowering therapy [LDL<1.4mmol/l] and decreased by 50% compared to the baseline).
  Interventions: Drug: OMT strategy

INTERVENTIONS:
Procedure: PCI strategy — -In the intervention group, vulnerable plaque lesions (quantitative flow ratio, QFR >0.8) to be treated at the operator's discretion using second-generation drug eluting stent (DES).
  Arms: PCI+OMT
Drug: OMT strategy — * Lifestyle modifications and intensive medical therapy (based on current guideline-directed secondary prevention).
  * Both groups to receive statin or other therapies to achieve LDL-C <1.4 mmol/L and decrease by 50% compared to the baseline.
  * Lifestyle and risk factor management to include smoking cessation, nutritional optimization, physical activity, adherence to prescribed medications, and control of diabetes and hypertension.

SUMMARY:
The aim of this clinical trial is to explore the optimal preventative treatment strategy for non-flow-limiting vulnerable plaques. The main question it aims to answer is:

Can interventional therapy further improve the outcome of non-flow-limiting vulnerable plaques on top of optimal pharmacologic therapy?

Researchers will randomly assign patients who meet the inclusion criteria to preventative intervention plus optimal drug therapy (experimental group) or optimal drug therapy alone (control group).

Participants will:

Assigned to the control group: optimized drug therapy consisting of lifestyle improvement and intensive drug therapy including high-dose statin or other therapy to achieve target levels (low-density lipoprotein cholesterol <1.4 mmol/L and decreased by 50% compared to the baseline). Lifestyle improvement and risk factor management included smoking cessation, nutritional optimization, physical activity, compliance with prescribed medications, and control of diabetes and hypertension.

Assigned to the experimental group: all non-flow-limiting vulnerable plaques were treated with conventional second-generation drug-eluting stents. After the procedure, participants received dual antiplatelet therapy for about 12 months as well as other medications in the control group.

ELIGIBILITY:
Inclusion Criteria Clinical Inclusion Criteria 1. Males or non-pregnant females aged 18-80 years 2. Clinically diagnosed with acute coronary syndrome (including unstable angina, ST-segment elevation myocardial infarction, and non-ST-segment elevation myocardial infarction) 3. Patients willing and able to sign a written informed consent form Angiography, QFR, and OCT Inclusion Criteria

1. Successful completion of angiography, QFR, and OCT examinations
2. Successful treatment of all culprit lesions and flow-limited lesions (QFR ≤ 0.8)
3. Reference vessel diameter between 2.5-4.0 mm on imaging assessment
4. Lesion length ≤40 mm
5. At least one significant stenosis (diameter reduction >50%) demonstrated by angiography, with QFR >0.80 and OCT-defined TCFA (fibrous cap thickness <65μm, lipid arc >90°)

Exclusion Criteria Clinical Exclusion Criteria

1. Patients with contraindications to dual antiplatelet therapy (DAPT) or planning to discontinue DAPT within one year
2. Patients with other major illnesses and a life expectancy <2 years
3. Patients scheduled for cardiac surgery or major non-cardiac surgery
4. Women who are breastfeeding, pregnant, or planning pregnancy during the study
5. Patients with severe heart failure (NYHA class III-IV or Killip class III-IV or left ventricular ejection fraction <35%)
6. Patients with estimated glomerular filtration rate <30 mL/(min·1.73 m²)
7. Patients with allergy to contrast agents or DES drugs
8. Patients currently enrolled in other clinical studies Angiographic Exclusion Criteria

1. Patients for whom CABG is the preferred treatment 2. Target lesion is a previously stented lesion 3. Target lesion is a post-bypass lesion 4. Target lesion is a heavily calcified or angulated lesion 5. Target lesion requires dual-stent technique 6. Target lesion is a left main coronary artery lesion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2190 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure | From enrollment to the end of treatment at 24 months
  Composite endpoint of cardiac death, target vessel myocardial infarction, ischemia-driven target vessel revascularization, and hospitalization for unstable or worsening angina.

SECONDARY OUTCOMES:
Death | From enrollment to the end of treatment at 24 months
  Including all-cause mortality, cardiovascular mortality, or non-cardiovascular mortality. All-cause mortality: Deaths classified as cardiac, non-cardiac, or of unknown cause. Cardiovascular mortality: Deaths due to direct cardiac causes (e.g., acute myocardial infarction, congestive heart failure, fatal arrhythmia), sudden cardiac death, and all deaths related to surgery or concomitant treatment. Non-cardiovascular mortality: Deaths definitively attributed to non-cardiac disease.
Myocardial infarction | From enrollment to the end of treatment at 24 months
  Including spontaneous myocardial infarction, perioperative myocardial infarction, and target vessel or non-target vessel-related myocardial infarction. Myocardial infarction: Based on the Fourth Edition Global Myocardial Infarction Definition Criteria. Spontaneous myocardial infarction: Includes types 1, 2, 4b, and 4c in the Fourth Edition Global Myocardial Infarction Classification. Perioperative myocardial infarction: Includes types 4a and 5 in the fourth edition of the Global Myocardial Infarction Classification. Target vessel myocardial infarction: Refers to ischemic necrosis of myocardial tissue supplied by the target vessel where a stent was implanted, resulting from in-stent thrombosis, restenosis, or other causes following coronary intervention. Non-target vessel myocardial infarction: Refers to ischemic necrosis in the corresponding myocardial region following coronary intervention due to obstruction or spasm in a non-target vessel.
Revascularization | From enrollment to the end of treatment at 24 months
  Revascularization refers to repeat percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG). All revascularization events will be classified as either ischemia-driven or non-ischemia-driven. A revascularization will be considered ischemia-driven if, upon coronary angiography, the re-implanted coronary segment exhibits ≥50% diameter stenosis and meets any one of the following ischemia-related criteria: a) History of chest pain (potentially related to the target vessel) b) Electrocardiographic changes at rest or objective evidence of ischemia during exercise testing or equivalent conditions (potentially related to the target vessel) c) Abnormal results from any invasive functional diagnostic test such as FFR
Hospitalization for any cause | From enrollment to the end of treatment at 24 months
  Hospitalization for any cause: Refers to a patient being admitted to an inpatient ward or emergency department with a minimum hospital stay of 24 hours. Additionally, the reason for readmission will be classified based on any cause, cardiac cause, or non-cardiac cause.
Intrastent thrombus | From enrollment to the end of treatment at 24 months
  Intrastent thrombus: Defined according to the explicit or probable criteria established by the Academic Research Consortium (ARC).
Stroke | From enrollment to the end of treatment at 24 months
  Stroke: Refers to the sudden onset of neurological dysfunction caused by impaired cerebral blood flow or intracerebral hemorrhage, in the absence of obvious non-vascular causes such as trauma, tumors, or infections.
Bleeding events | From enrollment to the end of treatment at 24 months
  Bleeding events: Events are assessed according to the Bleeding Academic Research Consortium (BARC) criteria. Severe bleeding is defined as BARC grades 3-5.
Major adverse cardiovascular events | From enrollment to the end of treatment at 24 months
  Major adverse cardiovascular events: cardiovascular death, non-fatal myocardial infarction, or unplanned rehospitalization due to unstable or progressive angina.
Patient-oriented outcomes | From enrollment to the end of treatment at 24 months
  Patient-oriented outcomes: A composite endpoint comprising death from any cause, myocardial infarction, or repeat revascularization.
Angina symptoms | From enrollment to the end of treatment at 24 months
  Angina symptoms: Based on the Seattle Angina Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables,figures, and appendices).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.